CLINICAL TRIAL: NCT05066672
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of NV-5138 in Adults With Treatment Resistant Depression
Brief Title: Phase 2 Study of NV-5138 in Adults With Treatment Resistant Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Navitor Pharmaceuticals, Inc. (Industry)
Collaborators: Supernus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NAV-17A-007; SPN820 (Other: Supernus Pharmaceuticals, Inc.)
Record Dates: First submitted 2021-09-23; First posted 2021-10-04 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — NV-5138

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, placebo-controlled
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: matched placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NV-5138 400 mg oral capsules (Experimental): Either 2 or 4 400 mg oral capsules administered once daily
  Interventions: Drug: NV-5138
- matched placebo (Placebo Comparator): 2 or 4 oral capsules administered once daily
  Interventions: Drug: matched placebo

INTERVENTIONS:
Drug: NV-5138 — NV-5138 is a novel, orally bioavailable, selective, direct activator of mTORC1 cellular signaling
  Other Names: SPN820
  Arms: NV-5138 400 mg oral capsules
Drug: matched placebo — matched placebo oral capsules
  Other Names: placebo; PBO
  Arms: matched placebo

SUMMARY:
This study will evaluate the efficacy and safety of NV-5138 in adults with TRD

DETAILED DESCRIPTION:
The is a multicenter, randomized, double-blind, flexible- dose, placebo-controlled, parallel design of adjunctive NV-5138 in adults with TRD.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18 to 70 years at Screening.
* Diagnosis of Major Depressive Disorder (MDD) according to the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) for either recurrent or single episode MDD without psychotic features that is confirmed by the Mini International Neuropsychiatric Interview (MINI).
* Montgomery-Asberg Depression Rating Scale (MADRS) Total Score of ≥26 for the current MDE at all Screening visits and Baseline (Day 1).
* CGI-S score of ≥4 (moderately ill or worse) at all Screening visits and Baseline.
* History of inadequate response to ≥2 but ≤4 prior ADT therapies (including the current ADT for the current MDE) ≥ 2 weeks at Screening and ≥ 8 weeks at Baseline.
* Stable therapeutic dose of one of the following ADTs for the current MDE for ≥2 weeks prior to Screening and maintain the therapeutic dose throughout the study: citalopram, escitalopram, paroxetine, fluoxetine, sertraline, duloxetine, venlafaxine (IR or XR), desvenlafaxine, or vortioxetine.
* Detectable blood level of the approved ADT at Visits 1 and 2 of the Screening Period.

Exclusion Criteria:

* MADRS Total Score improvement of ≥25% from the highest to the lowest score at any visit during the Screening Period.
* Clinically significant abnormal laboratory profiles, vital signs, or electrocardiograms (ECGs), per Investigator judgment.
* Judged by the Investigator to be at significant risk for suicide, violence, or homicide; or answers 'Yes' to items 4 or 5 on the Suicidal Ideation section of the C-SSRS at Screening or at Baseline; or has attempted suicide within the 6 months prior to Screening.
* History of psychotic disorder, including but not limited to schizophrenia, MDD with psychotic features, or bipolar I/II disorder with psychotic features.
* History of PTSD, OCD, panic disorder, intellectual disability, autism, acute stress disorder, or Cluster A or B personality disorder (per DSM-5 criteria).
* Any condition or procedure that may interfere with the absorption, metabolism, or elimination of the study medication (e.g., cholecystectomy or gastric bypass).
* In the Investigator's opinion, is unlikely to comply with the protocol or is unsuitable for any other reason.
* History of alcohol and/or substance use disorder within 6 months prior to Screening or is currently using or has positive results at Screening for drugs of abuse or has a positive alcohol result at any Screening or Baseline visit.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2025-02-15 (Actual); Study Completion 2025-02-15 (Actual)

PRIMARY OUTCOMES:
Evaluation of the efficacy of NV-5138 as measured by the Montgomery-Asberg Depression Rating scale | 5 weeks
  Change from Baseline to end of treatment period on the Montgomery-Asberg Depression Rating Scale (MADRS) Total Score. MADRS captures a clinician-rated score on a seven-point Likert scale for a score ranging from 0 to 60, with higher scores reflecting greater depression severity.

SECONDARY OUTCOMES:
Evaluation of the efficacy as measured by Clinical Global Impression-Severity (CGI-s) score | 5 weeks
  Change from baseline to end of treatment period on the Clinical Global Impression-Severity score for NV-5138 treated patients as compared to placebo. The CGI-S is a clinican-rated seven point scale from 0-7 where a higher rating represents higher severity of illness.

CONTACTS AND LOCATIONS:
Overall Officials: Randy Owen, MD, Study Director — Medical Monitor
Locations (1):
- Northwest Clinical Research Center, Inc., Bellevue, Washington, United States

IPD SHARING:
Plan to Share IPD: No